CLINICAL TRIAL: NCT06012071
Title: Comparison of Two-piece Zirconia Implants With Tissue-level and Bone-level Platform: Randomized Controlled Clinical Trial
Brief Title: Two-piece Zirconia Implants With Two Various Platforms
Acronym: ZircImpl
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZIRCIMPL001
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Edentulous Alveolar Ridge
Keywords: dental implants; zirconia; two-piece

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tissue-level (Active Comparator): Two-piece zirconia implants with tissue-level platform will be supplied to the single gap premolar regions in maxillae.
  Interventions: Device: Zirconia dental implants
- Bone-level (Experimental): Two-piece zirconia implants with bone-level platforms will be supplied to the single gap premolar regions in maxillae.
  Interventions: Device: Zirconia dental implants

INTERVENTIONS:
Device: Zirconia dental implants — Dental implants produced from zirconia material, either wit tissue-level or bone-level platform.

SUMMARY:
24 patients with missing premolar teeth and healed sockets will be recruited. They will be randomized into two groups to supplied with tissue-level (n=12) or bone-level (n=12) 10-mm long 4-mm wide zirconia implants. Primary and secondary stabilities will be measured with International Stability Quotient (ISQ) device. After 3 months, ceramic crowns will be supplied. Implant survival rates and parameters in relation to periimplant soft-tissues and bone health and anatomy will be recorded and evaluated after 1, 3 and 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Single missing maxillary premolar
* Occlusal stability
* Good oral hygiene
* Good general health

Exclusion Criteria:

* Oral mucosa pathology
* Dental caries
* Active periodontitis (non-treated)
* Systemic diseases and conditions that affect healing or immune capacity

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-07-03 (Actual); Primary Completion 2025-07-03 (Estimated); Study Completion 2027-12-03 (Estimated)

PRIMARY OUTCOMES:
Crestal bone loss (mm) | baseline, 1-year, 3-years, 5 years
  Loss of marginal bone in mm

SECONDARY OUTCOMES:
Probing depth (mm) | baseline, 1-year, 3-years, 5 years
  Probing pocket depth measured with periodontal probe
Bleeding on probing (BOP) | baseline, 1-year, 3-years, 5 years
  Bleeding provoked by probing
Volumetric tissue change | 1-year, 3-years, 5 years
  Sequential intraoral scanning

CONTACTS AND LOCATIONS:
Overall Officials: Rok Gašperšič, PhD, Principal Investigator — faculty of medicine
Locations (1):
- University Medical Centre, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No